CLINICAL TRIAL: NCT04928040
Title: Evaluation of Intracranial Pressure Change by Measuring Optic Nerve Sheath Diameter During Fluid Challenge
Brief Title: Effect of Fluid Challenge on Intracranial Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ozgur Komurcu, Assistant professor, Ondokuz Mayıs University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/436
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Fluid Challenge; Increased Intracranial Pressure
Keywords: optic nerve sheath diameter, fluid challenge
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluid challenge (Experimental): Fluid challenge effects on optic nerve sheath diameter
  Interventions: Diagnostic Test: Measurement of optic nerve sheath diameter

INTERVENTIONS:
Diagnostic Test: Measurement of optic nerve sheath diameter — The fluid challenge effects of optic nerve sheath diameter

SUMMARY:
Fluid challenge is frequently used in fluid management of critically ill patients. Assessing whether there is a preload reserve that can be used to increase the stroke volume by delivering a small amount of fluid in a short period of time. Optimization of fluid therapy is very important in intensive care patients. Inappropriate fluid therapy can cause significant morbidity and even mortality. Increased intracranial pressure is one of these important complications. In the present study, we planned to evaluate the effect of a fluid challenge on intracranial pressure by measuring the optic nerve sheath diameter (ONSD).

DETAILED DESCRIPTION:
The fluid challenge is a simple volume resuscitation evaluation method that provides an indication of the patient's likelihood of benefiting from an increase in the intravenous fluid volume. Both the fluid challenge and fluid responsiveness are evaluated by interpreting the change in hemodynamic parameters after 500 mL of crystalloid (or 250 mL of colloid) solution is infused over 10-15 min. This is done in an attempt to regulate the fluid therapy of hemodynamically unstable patients in order to prevent fluid overload. In the present study, we aim to investigate the effect of the fluid challenge maneuver on intracranial pressure in ICU patients with hemodynamic instability through measuring the optic nerve sheath diameter by ultrasonography.

Patients in the intensive care unit undergoing a fluid challenge were included in this prospective observational study. A fluid challenge is defined as a 500 mL crystalloid infusion administered over 10 min, and fluid responsiveness is defined as a subsequent increase in stroke volume of at least 15%. The ONSD and hemodynamic variables will be measured by ultrasonography before (T0), at the end (T1), and 30 min after the fluid challenge (T2). The primary outcome of the study is the change in intracranial pressure associated with the fluid challenge, and the secondary outcome is the relationship between fluid responsiveness and the change in ONSD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with no known intracranial pathology.
2. Patients with systolic blood pressure < 90 mmHg
3. Patients with mean blood pressure < 65 mmHg
4. Patients with tachycardia (heart rate 100 beats/min)
5. Patients with mottled skin, oliguria (diuresis of less than 20 ml/hr or 0.5 ml/kg/hr for two hours), and acute renal failure.
6. Patients with arterial lactate concentration > 2 mmol/L

Exclusion Criteria:

1. Patients with known intracranial hypertension
2. Patients in the early postpartum period
3. Patients with severe mitral or aortic regurgitation
4. Patients with cardiac arrhythmia
5. Patients unable to be evaluated due to poor echogenicity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
The change in intracranial pressure associated with the fluid challenge | Before, at the end, and 30 min after the fluid challenge.
  The change in intracranial pressure according to the optic nerve sheath diameter measurements.

SECONDARY OUTCOMES:
The relationship between fluid responsiveness and the change in optic nerve sheath diameter | Before, at the end, and 30 min after the fluid challenge.
  The fluid responsiveness associated with the change in optic nerve sheath diameter measurements

CONTACTS AND LOCATIONS:
Overall Officials: ozgur komurcu, 1, Principal Investigator — zgrkom@gmail.com
Locations (1):
- Ondokuz Mayıs Universitesi, Atakent, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Primary and secondary study outcomes

REFERENCES:
- [Background] Hoste EA, Maitland K, Brudney CS, Mehta R, Vincent JL, Yates D, Kellum JA, Mythen MG, Shaw AD; ADQI XII Investigators Group. Four phases of intravenous fluid therapy: a conceptual model. Br J Anaesth. 2014 Nov;113(5):740-7. doi: 10.1093/bja/aeu300. Epub 2014 Sep 9. PMID 25204700
- [Background] Cecconi M, Parsons AK, Rhodes A. What is a fluid challenge? Curr Opin Crit Care. 2011 Jun;17(3):290-5. doi: 10.1097/MCC.0b013e32834699cd. PMID 21508838
- [Background] Rajajee V, Vanaman M, Fletcher JJ, Jacobs TL. Optic nerve ultrasound for the detection of raised intracranial pressure. Neurocrit Care. 2011 Dec;15(3):506-15. doi: 10.1007/s12028-011-9606-8. PMID 21769456
- [Background] McGuire G, Crossley D, Richards J, Wong D. Effects of varying levels of positive end-expiratory pressure on intracranial pressure and cerebral perfusion pressure. Crit Care Med. 1997 Jun;25(6):1059-62. doi: 10.1097/00003246-199706000-00025. PMID 9201061
- [Derived] Komurcu O, Cicek E, Akyurt D, Kusderci HS, Dogru S, Koc K, Suren M. Reliability and validity of the Turkish form of intensive care nursing activities score. BMC Nurs. 2024 Nov 6;23(1):810. doi: 10.1186/s12912-024-02490-y. PMID 39506784